CLINICAL TRIAL: NCT02537951
Title: Autofluorescent Flavoprotein Imaging of Intraepidermal Nerve Fibers: a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Joost LM Jongen, Dr. J.L.M. Jongen, neurologist, Erasmus Medical Center
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: NL49568.078.14
Record Dates: First submitted 2015-08-22; First posted 2015-09-02 (Estimated); Results first posted 2019-06-03 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-02

CONDITIONS: Small Fiber Neuropathy
Keywords: autofluorescent flavoprotein imaging, capsaicin
MeSH Terms: conditions — Small Fiber Neuropathy

STUDY DESIGN:
Intervention Model Description: subjects are first undergoing measurements of AFI intensities following increasing nociceptive stimulus intensities, consequently it is tested whether the AFI activity can be blocked by lidocaine/prilocaine and a 8% capsaicin patch, i.e. whether the AFI activity is specific for nociceptor-acitivity
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- AFI intensity in healthy volunteers (Experimental): 10 healthy volunteers, on whose 3rd fingertips AFI intensity is measured through an AFI microscope
  Interventions: Device: AFI microscope
- negative control 1: lidocaine/prilocaine (Active Comparator): 10 healthy volunteers, on whose 3rd fingertips AFI intensity is measured through an AFI microscope, 1hour after application of lidocaine/prilocaine creme (negative control 1)
  Interventions: Device: negative control 1: lidocaine/prilocaine
- negative control 2: 8% capsaicin (Active Comparator): -10 healthy volunteers, on whose 3rd fingertips AFI intensity is measured through an AFI microscope, 1week after application of an 8% capsaicin patch (negative control 2)
  Interventions: Device: negative control 2: 8% capsaicin

INTERVENTIONS:
Device: AFI microscope — measurement of AFI intensities following increasing nociceptive stimulus intensities
  Arms: AFI intensity in healthy volunteers
Device: negative control 1: lidocaine/prilocaine — measurement of AFI intensities following lidocaine/prilocaine cream
  Arms: negative control 1: lidocaine/prilocaine
Device: negative control 2: 8% capsaicin — measurement of AFI intensities following 8% capsaicin patch
  Arms: negative control 2: 8% capsaicin

SUMMARY:
Small fiber neuropathy (SFN) is a common disorder, which has a profound negative impact on quality of life because of severe neuropathic pain. To reliably establish a diagnosis of SFN is challenging, since neurological examination and nerve conduction studies are often normal. Autofluorescent flavoprotein imaging (AFI) is an optical method through which neuronal activity in the termination area of small nerve fibers in the spinal cord can be quantified. Since the epidermis also contains a high density of small nerve terminals and since the number of intraepidermal nerve fibers is greatly reduced in patients with SFN, our hypothesis is that AFI intensity is reduced in patients with SFN. To support this hypothesis, a pilot study is required in which the investigators first need to confirm the precision of AFI in the epidermis of the third finger of 10 healthy volunteers. Secondly, lidocaine/prilocaine cream will be used as a negative control. Finally, the AFI signal will be measured after application of a 8% capsaicin patch, through which (temporarily) a selective reduction of small nerve fibers can be induced, mimicking SFN. Using this experimental design, the investigators will be able to test the reliability and validity of AFI for capsaicin-induced small nerve fiber degeneration. This would be a significant step in developing an objective, rapid and non-invasive diagnostic tool to diagnose patients with SFN, which may also be utilized as a biomarker in studies that assess the efficacy of novel treatments for SFN.

DETAILED DESCRIPTION:
The first aim of the current project is to test the precision of AFI in the epidermis of 10 healthy volunteers. For this purpose, a range of nociceptive electrical stimuli with increasing intensities (5Hz @ 0.5mA-1.0mA) and one innocuous control stimulus (2000Hz @1mA) will be delivered to the third finger of each subject. The outcome measure is AFI-intensity, which is the change in autofluorescence intensity compared to baseline (delta F/F). The standard deviation of AFI intensity will be the measure of precision. Pearson's correlation coefficient will be calculated between electrical stimulus intensities and AFI intensity. A linear correlation needs to be confirmed, since this is a general characteristic of AFI. A paired t-tests will be performed to compare AFI intensities following 5Hz @ 1mA stimulation and 2000Hz @ 1mA stimulation. Lidocaine/prilocaine cream will be applied to the fingertips of the subjects and the electrical stimuli will be repeated, to serve as a negative control experiment. A repeated-measures ANOVA will be performed to compare AFI intensities before and after application of lidocaine/prilocaine cream.

The second aim of our study is to validate AFI in experimentally induced small nerve fiber degeneration of the epidermis, by comparing AFI intensities in subjects before and one week after application of a 8% capsaicin patch to the third fingertip. A repeated-measures ANOVA will be performed to compare AFI intensities before and after capsaicin-induced small nerve fiber degeneration. Assuming that all subjects develop epidermal small fiber degeneration following the 8% capsaicin patch, a statistically significant difference in AFI intensity would serve as a proof-of-principle and would provide validity to autofluorescent flavoprotein imaging of epidermal nociceptor activity as a diagnostic test for SFN. Comparing the distributions of before and after capsaicin-induced small nerve fiber degeneration will lead to a probability estimation of having SFN based on the outcome measure, i.e. AFI intensity. In future research, false-positive and false-negative consequences will be evaluated, leading to cut-off values in patients suspected for SFN.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers

Exclusion Criteria:

* younger than 18 years
* pre-existing neuropathy
* previous allergic reaction to local anaesthetics

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-09; Primary Completion 2016-07 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joost LM Jongen, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Dept. Neurology, Erasmus MC, Rotterdam, Netherlands

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: all 10 healthy volunteers underwent 3 experiments, all 10 have completed these experiments:
  1. AFI intensity measurements
  2. lidocaine/prilocaine creme, one hour later followed by AFI intensity measurements
  3. capsaicin patch (2 hours after lidocaine/prilocaine creme), one week later followed by AFI intensity measurements
Groups:
- 10 Healthy Volunteers: 10 healthy volunteers underwent three procedures, always in the same order:
  1. baseline AFI measurements
  2. application of lidocaine/prilocaine creme, 1 hour later followed by AFI measurements
  3. application of capsaicin patches, 1 week later followed by AFI measurements
Period: Overall Study
Arm/Group | 10 Healthy Volunteers
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- AFI Intensity in Healthy Volunteers: 10 healthy volunteers, on whose 3rd fingertips AFI intensity is measured through an AFI microscope
  AFI microscope: measurement of AFI intensities following increasing nociceptive stimulus intensities
  After AFI intensity measurements, the same experiment will be repeated one hour after application of lidocaine/prilocaine creme
  After the negative control experiment using lidocaine/prilocaine creme, AFI intensity measurements will be repeated one week after application of a capsaicin 8% patch (second negative control experiment)
Arm/Group | AFI Intensity in Healthy Volunteers
Number analyzed (Participants) | 10
Age, Continuous [Median (Full Range); unit: years] | 25 [20 to 30]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Netherlands | 10

OUTCOME MEASURES:

1. Primary Outcome: AFI-intensity After Nociceptive Stimulation
Description: AFI-intensity (delta F/F) at the 3rd fingertip, directly after application of grading nociceptive stimuli
Time Frame: Day 1, T=0h (AFI measurements), Day 1, T=6h (AFI measurements after lidocaine/prilocaine), Day 7 (AFI measurements after capsaicin)
Measure: Mean (Standard Error); unit: unitless
Arm/Group | AFI Intensity in Healthy Volunteers | Negative Control 1: Lidocaine/Prilocaine | Negative Control 2: 8% Capsaicin
Number analyzed (Participants) | 10 | 10 | 10
unitless | 0.60 (0.25) | 0.25 (0.25) | 0.50 (0.50)

ADVERSE EVENTS:
Time Frame: 1 month
Groups:
- AFI Intensity in Healthy Volunteers: 10 healthy volunteers-AFI intensity measurements
- Negative Control 1: Lidocaine/Prilocaine: 10 healthy volunteers-lidocaine/prilocaine creme, one hour lat
- Negative Control 2: 8% Capsaicin: 10 healthy volunteers-capsaicin patch (2 hours after lidocaine
Arm/Group | AFI Intensity in Healthy Volunteers | Negative Control 1: Lidocaine/Prilocaine | Negative Control 2: 8% Capsaicin
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2014-06-23): https://cdn.clinicaltrials.gov/large-docs/51/NCT02537951/Prot_000.pdf